CLINICAL TRIAL: NCT04698005
Title: Exogenous Ketones for Acutely Decompensated Heart Failure
Acronym: KADHEF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Marek Sramko, Head of the Department of Acute Cardiology, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-20-28
Record Dates: First submitted 2020-12-02; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Acute Heart Failure; Low Cardiac Output Syndrome; Hemodynamic Instability; Ketosis
MeSH Terms: conditions — Cardiac Output, Low; Ketosis

STUDY DESIGN:
Intervention Model Description: randomisation 1:1 to active treatment (exogenous ketones) vs. placebo (drinking water of equivalent volume)
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participant and the physician in charge of the participant will be blinded to the given treatment (ketone drink vs. placebo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Supplementation of exogenous ketones (Experimental): Exogeneous ketones will be administered orally using monoester 3-OHB concentrate without added salts (25g 3-OHB in 65ml H.V.M.N Ketone Ester, H.V.M.N, USA or equivalent). The drink will be administered over 10 mins every 3 hours, 3 times in a row.
  Interventions: Dietary Supplement: 25g Ketone monoester without added salts
- Control group (Placebo Comparator): The patients will receive a placebo drink (drinking water) of equivalent volume (3x 65ml)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 25g Ketone monoester without added salts — oral supplementation of ketone monoester
  Other Names: 25g 3-OHB in 65ml, H.V.M.N Ketone Ester, H.V.M.N, USA or equivalent
  Arms: Supplementation of exogenous ketones
Other: Placebo — The patients will receive a placebo drink (drinking water) of equivalent volume (3x 65ml)
  Arms: Control group

SUMMARY:
This study will evaluate whether supplementation of exogenous ketones in patients with severe left ventricular dysfunction and acutely decompensated heart failure requiring inotropic therapy would improve the patient's hemodynamics and symptoms.

DETAILED DESCRIPTION:
The study will include patients with acutely decompensated chronic heart failure requiring inotropic therapy for the syndrome of low cardiac output. While being on the inotropic therapy, the patients will be randomized to oral supplementation of exogenous ketones vs. placebo, which will be repeatedly administered over 9 hours. The patients will undergo continuous invasive hemodynamic monitoring by pulmonary artery catheter, repeated laboratory assessment, and repeated assessment of the severity of symptoms for 24 hours.

Exogenous ketones will be administered orally using monoester 3-OHB concentrate without added salts (25g 3-OHB in 65ml H.V.M.N Ketone Ester, H.V.M.N, USA or equivalent). The drink will be administered over 10 mins every 3 hours, 3 times in a row (hour 0, 3, 6).

All patients with K<3.7 mmol/l will receive a continuous infusion of 7.5% potassium until reach target K levels of 4.0-4.9 mmol /l. Glycemia will be controlled as needed by insulin and dextrose to maintain glucose concentration of 4 - 12 mmol/l

All patients will receive standard treatment of acute heart failure, including intravenous diuretics and inotropic therapy. The recommended inotropic therapy will include milrinone 0.5 ug/kg/min, levosimendan 0.1 ug/kg/min up to 25mg without initial bolus, or dobutamine 0.5 ug/kg/min in patients without chronic therapy with beta-blockers.

The severity of symptoms will be self-reported by the patient using 1-10 visual analog scale.

Workflow:

* Hemodynamic assessment, assessment of ketones concentration: 1-3h before randomization, 0-9h hourly, 16-24h (next morning)
* Biochemical assessment (renal function, liver enzymes, BNP, hs-TnT) 0h, 9h, 16-24h
* Assessment of symptoms and Scv02: 0h, 1h, 3h, 9h, 16-24h

Statistical methods:

Each study arm will include 12 patients. The study size was estimated to have power of (1 - beta) of 0.8 and alpha of 5% for between-group comparison of changes in cardiac index and stroke volume index by ANOVA and for comparison of the changes in cardiac index and stroke volume index by paired t-tests.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure due ischemic or nonischemic cardiomyopathy
* Acute decompensation of heart failure with the need of inotropes
* Achievement of relative stabilization on inotropes (INTERMACS class >2)
* Left ventricular ejection fraction <= 35%
* Age >18 years

Exclusion Criteria:

* Deteriorating cardiogenic shock with likely need of mechanical circulatory support in the subsequent 48 hours
* Chronic kidney disease grade 4 or 5
* Diabetic ketoacidosis (3-OHB >2mmol/l at baseline)
* Hemodynamic severe arrhythmias
* Acute heart failure due to transient triggers (acute coronary syndrome, atrial fibrillation, infection etc..)
* Contraindications to invasive hemodynamic monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum change of stroke volume index | Maximum value of stroke volume index measured between hour 1 - 3 of the study protocol at 15-minute intervals
  Maximum change of stroke volume index (ml/m2) between baseline and hour 1 - 3
Maximum change of cardiac index | Maximum value of cardiac index measured between hour 1 - 3 of the study protocol at 15-minute intervals
  Maximum change of cardiac index (L/m2) between baseline and hour 1 - 3
Change of mean stroke volume index | Mean value of stroke volume index measured every 15 minutes during 9 hours of the study protocol
  Difference between baseline stroke volume index and mean stroke volume index (ml/m2) during the study protocol
Change of mean cardiac index | Mean value of cardiac index measured every 15 minutes during 9 hours of the study protocol
  Difference between baseline cardiac index (L/m2) and mean cardiac index during the study protocol

SECONDARY OUTCOMES:
Change in patient/symptoms | Symptoms scored at hours 0, 1, 10, 24 and expressed as an area under the curve
  Change in patient-referred symptoms by visual-analog scale (1=unbearable dyspnea, 10=no symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided